CLINICAL TRIAL: NCT05155995
Title: A Randomized, Open Label, Single Dose, 2-way Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety Between After Administration of a Fixed-dose Combination Drug of HCP2001 and Co-administration of Each Component in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HCP2001 and Co-administration of Each Component in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-DATAM-101
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Period 1: Fasted state + RLD2007 +RLD2008 + RLD2102
  Period 2: Fasted state + HCP2001
  Interventions: Drug: HCP2001; Drug: RLD2007; Drug: RLD2008; Drug: RLD2102
- Sequence 2 (Experimental): Period 1: Fasted state + HCP2001
  Period 2: Fasted state + RLD2007 +RLD2008 + RLD2102
  Interventions: Drug: HCP2001; Drug: RLD2007; Drug: RLD2008; Drug: RLD2102
- Sequence 3 (Experimental): Period 1: High fat diet + RLD2007 +RLD2008 + RLD2102
  Period 2: High fat diet + HCP2001
  Interventions: Drug: HCP2001; Drug: RLD2007; Drug: RLD2008; Drug: RLD2102
- Sequence 4 (Experimental): Period 1: High fat diet + HCP2001
  Period 2: High fat diet + RLD2007 +RLD2008 + RLD2102
  Interventions: Drug: HCP2001; Drug: RLD2007; Drug: RLD2008; Drug: RLD2102

INTERVENTIONS:
Drug: HCP2001 — Take it once per period.
Drug: RLD2007 — Take it once per period.
Drug: RLD2008 — Take it once per period.
Drug: RLD2102 — Take it once per period.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HCP2001 and co-administration of each component in fasting and fed conditions respectively in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers 19 kg/m^2 ≤ BMI < 28 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug.
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
AUCt | 0~48hr
  Pharmacokinetic evaluation
Cmax | 0~48hr
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~48hr
  Pharmacokinetic evaluation
Tmax | 0~48hr
  Pharmacokinetic evaluation
t1/2 | 0~48hr
  Pharmacokinetic evaluation
CL/F | 0~48hr
  Pharmacokinetic evaluation
Vd/F | 0~48hr
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mingeul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea